CLINICAL TRIAL: NCT04723849
Title: Efficacy Evaluation of a Mixed Compound (Magnesium, Curcumin, Resveratrol, Quercetin, Vitamin E, Zinc, Selenium, Folic Acid, Vitamin D) in Terms of Endothelium Damage/Function in Pediatric Subjects With Obesity: Double-blind, Randomized, Controlled Trial of 6-months Duration.
Brief Title: Efficacy Evaluation of a Mixed Compound of Antioxidants in Terms of Endothelium Damage/Function in Pediatric Subjects With Obesity.
Acronym: OBELIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Angelo Pietrobelli, Professor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 5384
Record Dates: First submitted 2021-01-14; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Using a computer-generated randomization schedule, study supplement and placebo were randomized (1:1) into 70 batches (each consisting of 6 packs containing 30 tablets a pack) and each was given a unique identification number. The coordinator of the study maintained the randomization list. Study physicians, other study personnel, and parents or legal guardians were blinded to of the batches of medication and to the identification. Subjects who satisfied the inclusion for the study were assigned an identification number (linked to a batch) in sequential order. Subjects took one tablet per day orally starting day one after the visit and continuing for the 6-month duration of the study. A number of tablets not taken equal to of greater of 2 tablets/month was considered not adherence to the study (drop out).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Using a computer-generated randomization schedule, study supplement and placebo were randomized (1:1) into 70 batches (each consisting of 6 packs containing 30 tablets a pack) and each was given a unique identification number. The coordinator of the study maintained the randomization list. Study physicians, other study personnel, and parents or legal guardians were blinded to of the batches of medication and to the identification. Subjects who satisfied the inclusion for the study were assigned an identification number (linked to a batch) in sequential order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tretment group (Experimental): Subjects took one tablet per day orally starting day one after the visit and continuing for the 6-month duration of the study.
  Interventions: Dietary Supplement: Auxilie® Immuplus, Envicon Medical, Verona, Italy
- Placebo group (Placebo Comparator): Subjects took one tablet per day orally starting day one after the visit and continuing for the 6-month duration of the study.
  Interventions: Dietary Supplement: Auxilie® Immuplus, Envicon Medical, Verona, Italy

INTERVENTIONS:
Dietary Supplement: Auxilie® Immuplus, Envicon Medical, Verona, Italy — Subjects took one tablet per day orally starting day one after the visit and continuing for the 6-month duration of the study. Height (cm) and weight (kg) were measured for each child at every visit. Endothelial function was assessed using two methodologies: a "post occlusive release hyperemic test" (PORH) and a "heat provocation test" (HPT).

SUMMARY:
The aim of our study was to test the effects on endothelium of a combination of curcumin, resveratrol, plus zinc, magnesium, selenium and Vitamin D in a cohort of pediatric subjects with obesity.

DETAILED DESCRIPTION:
The aim of our study was to test the effects on endothelium of a combination of curcumin, resveratrol, plus zinc, magnesium, selenium and Vitamin D in a cohort of pediatric subjects with obesity. Endothelial function was assessed using two methodologies: a "post occlusive release hyperemic test" (PORH) and a "heat provocation test" (HPT). Treatment tablet composition (Auxilie® Immuplus, Envicon Medical, Verona, Italy): Vitamin D3: 25,00 mcg, Folic acid: 90,00 mcg, Selenium: 55,00 mcg Magnesium: 300,00 mg, Zinc: 7,00 mg, Curcum (Meriva®): 100,00 mg Polygonum dry extract: 20,41 mg (of which Resveratrol: 20,00 mg), Soy dry extract: 37,50 mg. Placebo tablet composition: Saccharose, fructose, aroma, anti-agglomerate agents: fatty acids magnesium salts, silicium dioxide, colorant: riboflavin 5-sodium phosphate; sweetener: stevia glycoside, sucralose, neosperidin DC. Both tablets (treatment and placebo) were similar in form, color and flavor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of obesity as defined by a BMI higher than the 95 percentile for age based on the CDC standard
* Age 6-17 years

Exclusion Criteria:

* Children with genetic syndromes or cardiovascular diseases were excluded from the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
To test the effects on endothelium of a combination of curcumin, resveratrol, plus zinc, magnesium, selenium and Vitamin D in a cohort of pediatric subjects with obesity. | 6 months
  Endothelial function was assessed using a "post occlusive release hyperemic test". (PORH). Unit of measure: arbitrary perfusion units (PU)

SECONDARY OUTCOMES:
To test the effects on endothelium of a combination of curcumin, resveratrol, plus zinc, magnesium, selenium and Vitamin D in a cohort of pediatric subjects with obesity. | 6 months
  Endothelial function was assessed using "heat provocation test" (HPT). Unit of measure: arbitrary perfusion units (PU)

OTHER OUTCOMES:
To test the effects on endothelium and body composition of a combination of curcumin, resveratrol, plus zinc, magnesium, selenium and Vitamin D in a cohort of pediatric subjects with obesity. | 6 months
  Height (cm), Weight (kg) used to calculate BMI (Kg/m2)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: Undecided